CLINICAL TRIAL: NCT00258349
Title: A Phase I/II Study of Suberoylanilide Hydroxamic Acid (SAHA) in Combination With Trastuzumab (Herceptin) in Patients With Advanced Metastatic and/or Local Chest Wall Recurrent Her-2 Amplified Breast Cancer
Brief Title: Vorinostat and Trastuzumab in Treating Patients With Metastatic or Locally Recurrent Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00503; NCI-2009-00503 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000449963; E1104 (Other: Eastern Cooperative Oncology Group); E1104 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Vorinostat; Trastuzumab

ARMS (1):
- Arm I (Experimental): Patients will receive vorinostat by mouth twice a day for 2 weeks. They will also receive a 90-minute infusion of trastuzumab in week 1.
  Interventions: Drug: vorinostat; Drug: trastuzumab

INTERVENTIONS:
Drug: vorinostat — Given orally
Drug: trastuzumab — Given IV

SUMMARY:
This phase I/II trial is studying the side effects and best dose of vorinostat when given together with trastuzumab and to see how well they work in treating patients with metastatic breast canceror breast cancer that has recurred in the chest wall. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Vorinostat and trastuzumab also may stop the growth of tumor cells by blocking blood flow to the tumor. Giving vorinostat together with trastuzumab may be a better way to block tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of vorinostat in combination with trastuzumab (Herceptin) in patients with metastatic or local chest wall recurrent HER-2-amplified breast cancer. (Phase I) II. To determine the toxic effects of this regimen in these patients. (Phase I) III. To determine the response rate in patients treated with this regimen. (Phase II)

SECONDARY OBJECTIVE:

I. To determine the time to progression in patients treated with this regimen. (Phase II)

OUTLINE: This is an open-label, multicenter, dose-escalation study of vorinostat.

PHASE I: Patients receive oral vorinostat twice daily on days 1-14 and trastuzumab (Herceptin®) IV over 90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of vorinostat until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity. At least 6 patients are treated at the MTD.

PHASE II: Patients receive vorinostat at the MTD and trastuzumab as in phase I.

After completion of study treatment, patients are followed periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active or ongoing infection
* No history of allergic reaction to compounds of similar chemical or biologic composition to vorinostat or other agents used in study
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin; 1 week for capecitabine) and recovered
* More than 3 weeks since prior radiotherapy and recovered
* Recovered from prior therapy
* At least 2 weeks since prior valproic acid
* More than 4 weeks since prior investigational agents
* More than 4 weeks since prior lapatinib ditosylate
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Measurable disease, defined as >= 1 unidimensionally measurable lesion > 20 mm by conventional techniques or > 10 mm by spiral CT scan
* No other concurrent investigational agents
* Concurrent bisphosphonates allowed provided therapy was initiated prior to study treatment
* No other concurrent anticancer therapy
* Recurrent or progressive disease while receiving prior trastuzumab (Herceptin) (with or without chemotherapy) OR relapsed within 3 months of last dose of prior adjuvant trastuzumab for metastatic disease
* Histologically confirmed breast cancer
* Must overexpress HER-2 gene
* Metastatic or chest wall recurrent disease
* Site of measurable disease must not have been irradiated (except chest wall recurrence treated with adjuvant radiation therapy)
* No untreated brain metastases
* Previously treated brain metastasis responsive to radiotherapy and/or surgery allowed provided the brain is not the sole site of measurable disease
* ECOG 0-2
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9 g/dL
* AST and ALT =< 2 times upper limit of normal
* Bilirubin =< 1.5 mg/dL (3 mg/dL in the presence of Gilbert's disease provided direct bilirubin is normal)
* Creatinine =< 1.5 mg/dL
* LVEF normal by nuclear scan or echocardiogram
* No evidence of PR prolongation or AV block by EKG
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-08; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramona Swaby, Principal Investigator — Eastern Cooperative Oncology Group
Locations (25):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Eastern Cooperative Oncology Group, Boston, Massachusetts
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Saint Vincent's Hospital and Medical Center of New York, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The phase I portion of the study was activated on August 23, 2006, and completed on June 28, 2007. The phase II portion of the study then was activated, and suspended on October 4, 2007, terminated on August 27, 2009, with a final accrual of 16 patients by ECOG institutes.
Groups:
- Vorinostat +Trastuzumab: Trastuzumab: 6 mg/kg once on Day 1, infused over 90 minutes, every 3 weeks; Vorinostat: 200 mg of SAHA orally twice a day, daily for 14 days out of a 21-day cycle.
Period: Overall Study
Arm/Group | Vorinostat +Trastuzumab
Started | 16
HER2-positive by Central Review | 10
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat +Trastuzumab
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Tumor response is assessed by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0. Response included complete response (CR) and partial response (PR). CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: Tumor assessment was obtained at baseline, after 6 weeks (week 6 = last week of Cycle 2), and after every 4 cycles of therapy
Population: 10 eligible HER2-positive (by central review) patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Vorinostat +Trastuzumab: Trastuzumab: 6 mg/kg once on Day 1, infused over 90 minutes, every 3 weeks;
  Vorinostat 200 mg of SAHA orally twice a day, daily for 14 days out of a 21-day cycle
Arm/Group | Vorinostat +Trastuzumab
Number analyzed (Participants) | 10
percentage of participants | 0 [0 to 26]

2. Secondary Outcome: Time to Progression
Description: Tumor response is assessed by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0. Disease progression is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s). Time to progression is defined as time from registration to disease progression.
Time Frame: as for outcome 1
Population: 10 eligible HER2-positive (by central review) patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorinostat +Trastuzumab
Number analyzed (Participants) | 10
months | 1.5 [1.3 to 3.7]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from registration to death from any cause. Patients who were alive were censored as the last date of known alive.
Time Frame: Survival was assessed every 3 months for first 2 years from protocol entry, then every 6 months until 3 years from study entry
Population: 10 eligible HER2-positive (by central review) patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorinostat +Trastuzumab
Number analyzed (Participants) | 10
months | 9.3 [5.1 to 24.7]

ADVERSE EVENTS:
Time Frame: For Phase I, toxicity was assessed once a week during Cycle 1 and at the end of each cycle for Cycles 2 and all subsequent cycles. For Phase II, assess toxicity at the end of every cycle (1 cycle = 21 Days) and 30 days after after the end of treatment.
Groups:
- Vorinostat +Trastuzumab (Phase II): Trastuzumab: 6 mg/kg once on Day 1, infused over 90 minutes, every 3 weeks; Vorinostat 200 mg of SAHA orally twice a day, daily for 14 days out of a 21-day cycle
- Vorinostat +Trastuzumab (Phase I): phase I patients for identify maximum tolerated dose
Arm/Group | Vorinostat +Trastuzumab (Phase II) | Vorinostat +Trastuzumab (Phase I)
Serious Adverse Events (participants affected / at risk) | 2/9 | 2/7
Other Adverse Events (participants affected / at risk) | 8/9 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat +Trastuzumab (Phase II) (N=9) | Vorinostat +Trastuzumab (Phase I) (N=7)
Thrombocytopenia (Investigations) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat +Trastuzumab (Phase II) (N=9) | Vorinostat +Trastuzumab (Phase I) (N=7)
Anemia (Blood and lymphatic system disorders) | 3 | 2
Leukopenia (Investigations) | 2 | 1
Neutropenia (Investigations) | 0 | 1
Thrombocytopenia (Investigations) | 2 | 1
Hypotension (Vascular disorders) | 0 | 1
Fatigue (General disorders) | 3 | 3
Insomnia (Psychiatric disorders) | 0 | 1
Weight loss (Investigations) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Nail change (Skin and subcutaneous tissue disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2
Creatinine increased (Investigations) | 4 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1 | 0
Taste disturbance (Gastrointestinal disorders) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Alanine aminotransferase (ALT) increased (Investigations) | 2 | 0
Aspartate aminotransferase (AST) increased (Investigations) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less